CLINICAL TRIAL: NCT01749163
Title: Determining the Extra-pancreatic Effects of Incretin Hormones During Euglycemic and Hyperglycemic Pancreatic Clamps
Brief Title: Hyperglycemia and the Extra-pancreatic Effect of Incretins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Senior Researcher, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PancClamp
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Extra-pancreatic Incretin Effect; Glucose Effectiveness
MeSH Terms: interventions — Sodium Chloride; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Experimental): Saline will be coninfused during the pancreatic clamp
  Interventions: Biological: Saline
- GIP (Experimental): GIP will be infused intravenously during the pancreatic clamp at 1.5 pmol/kg/min
  Interventions: Biological: GIP
- GLP-1 (Experimental): GLP-1 will be infused intravenously during the pancreatic clamp at 0.5 pmol/kg/min
  Interventions: Biological: GLP-1

INTERVENTIONS:
Biological: Saline
  Arms: Control
Biological: GIP
  Arms: GIP
Biological: GLP-1
  Arms: GLP-1

SUMMARY:
Incretin hormones (GLP-1 and GIP) released from the intestine in response to meal ingestion augment insulin secretion from the pancreas to help maintain glycemic control. Studies in vitro and in vivo have shown that these incretin hormones also have functional effects in other tissues independent of the insulin secretory response. Both GLP-1 and GIP stimulate insulin secretion in a glucose-dependent manner, however the glucose-dependency of their extra-pancreatic effects has not been examined in vivo. By using pancreatic clamp methodology during euglycemic and hyperglycemic conditions we will test the hypothesis that extra-pancreatic effects of GLP-1 and GIP are glucose-dependent.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* BMI 18-30 kg/m2
* Male
* Normal glycemic control (fasting glucose <5.6 mM)

Exclusion Criteria:

* Evidence of chronic disease
* Smoking
* Active weight loss (>2 kg in previous 6 months)
* Treatment with drugs known to affect our outcome varaibles

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | up to 4 hours
  Pancreatic clamp will be performed including infusion of somatostatin and replacement of basal insulin, glucagon, and growth hormone. During pancreatic clamps, euglycemia (5 mM) will be maintained via exogenous glucose infusion for the first 2-hours, followed by hyperglycemia (+5 mM) for the final 2-hours. An infusion of the stable isotope [U13C]glucose will be performed to assess glucose kinetics. Expired air will be collected for the analysis of [U13C]glucose into 13CO2.
Lipid metabolism | up to 4 hours
  An infusion of the stable isotope [D5]glycerol will be performed to assess glycerol kinetics.

SECONDARY OUTCOMES:
Endothelial function | Baseline, 2 hours, and 4 hours
  Ultrasound Doppler will be used to examine lower and upper limb blood flow and flow-mediated dilation
Signaling | Baseline, 2 hours, and 4 hours
  Skeletal muscle (vastus lateralis) and subcutaneous abdominal adipose biopsies will be obtained under local anaesthetic by the Bergstrom needle technique. Intracellular signalling related to glucose and lipid metabolism will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas PJ Solomon, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Solomon TPJ, Carter S, Haus JM, Karstoft K, von Holstein-Rathlou S, Nielsen MS, Gillum MP. Plasma FGF21 concentrations are regulated by glucose independently of insulin and GLP-1 in lean, healthy humans. PeerJ. 2022 Jan 19;10:e12755. doi: 10.7717/peerj.12755. eCollection 2022. PMID 35111398